CLINICAL TRIAL: NCT01347632
Title: Prospective Evaluation of the Impact of Bacterial Vaginosis and Its Treatment on Mucosal Susceptibility to HIV-1 Infection and Endpoints of Cervico-Vaginal Safety
Brief Title: Study of How Bacterial Vaginosis and Its Treatment Affects Cervical and Vaginal Tissue
Acronym: CONRADBV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CONRAD (Other)
Collaborators: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Annie Thurman, Associate Professor of OBGYN, CONRAD
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: D11115
Record Dates: First submitted 2011-04-15; First posted 2011-05-04 (Estimated); Results first posted 2014-08-26 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-11

CONDITIONS: Bacterial Vaginosis; Vaginal Discharge
Keywords: Bacterial Vaginosis; Vaginal discharge; Vaginal infections
MeSH Terms: conditions — Vaginosis, Bacterial; Vaginal Discharge; Vaginitis | interventions — Metronidazole

STUDY DESIGN:
Intervention Model Description: Open Label
Masking Description: This is an open label study - there was no masking
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BV pre treatment (Other): Open Label Study. All participants had BV and took metronidazole 500 mg po BID for 7 days.
  Interventions: Drug: Metronidazole

INTERVENTIONS:
Drug: Metronidazole — All participants had BV at baseline. They all received metronidazole 500 mg po BID for 7 days
  Other Names: Flagyl

SUMMARY:
This is a research study to determine whether bacterial vaginosis (BV) changes the cervico-vaginal tissue (skin covering the cervix and vagina) and makes women at higher risk for getting HIV (Human Immunodeficiency Virus). Vaginal and cervical tissue biopsies from women with BV will be obtained and infected OUTSIDE the body (ex vivo) with HIV.

BV is a vaginal infection that develops when there is an imbalance in the normal bacteria found in a woman's vagina. It is the most common cause of vaginal discharge among women of child-bearing age. BV infections potentially harm the safety of the tissue surrounding the cervico-vaginal region. When the cervico-vaginal tissue is not well protected, the risk of acquiring HIV from an infected partner might increase significantly. Studies have shown that HIV is more common in women with BV than in women with normal vaginal bacteria.

Treatment of BV typically involves the use of antibiotics. Antibiotics kill harmful bacteria and provide a temporary relief from the symptoms caused by the infection. Women participating in this study will use the generic antibiotic metronidazole, also known as Flagyl. The Center for Disease Control and Prevention (CDC) recommends Flagyl for the treatment of BV.

The study will evaluate HIV infection and safety of cervico-vaginal tissue in women at 3 different time periods:

1. During a BV infection
2. Approximately 1 week after completing a 7-day course of metronidazole therapy
3. Approximately 1 month after completing the 7-day course of metronidazole therapy

You will not come in contact with HIV during this study - only your samples (after we have removed them from your vagina/cervix) come in contact with HIV.

DETAILED DESCRIPTION:
WHY ARE YOU BEING ASKED TO TAKE PART?

You are being asked to participate in this research project because you are a female between the ages of 18-50 and you think you might have a current BV infection; your menstrual cycle is regular and your last two periods were 21-35 days apart; you are willing comply with the procedures done at 3 study visits; and you are willing to take metronidazole for 7 days.

This study includes only people who voluntarily choose to take part. Please take your time to make your decision and feel free to ask any questions you might have.

WHAT ARE SOME IMPORTANT DETAILS ABOUT THIS STUDY?

Up to approximately 80 women are expected to take part in the study at this local site. There are no other study sites participating in the study. You will have three scheduled visits to the clinic. Your participation in the study will last for approximately 2 months.

WHEN SHOULD YOU NOT TAKE PART?

You should not take part in this study if you:

* Drink alcohol on a daily basis and are unwilling to abstain from alcohol while taking metronidazole.
* Have a known allergy to metronidazole.
* Have chronic immune suppression (including, but not limited to, chronic steroid use, chronic anti-fungal use, Diabetes Mellitus, organ transplant).
* Had an abnormal documented Pap smear in the past 12 months.
* Had your last Depo medroxyprogesterone acetate (DMPA) injection less than 3 months ago and you have not had 2 normal menses since then.
* Used any hormonal contraceptive method within the past 2 months.
* Used oral or vaginal antibiotics or anti-fungals in the last 14 days.
* Had surgery or biopsy of the vulva, vagina, or cervix within 30 days.
* Had a hysterectomy.
* Were pregnant within the past 3 months.
* Are currently breastfeeding.
* Are HIV-1 positive, or your current sexual partner(s) is.
* Use daily anti-viral suppression medications for Herpes Simplex Virus (HSV).
* Believe you currently have a sexually transmitted infection.
* Used a douche or other vaginal products or put anything in your vagina in the past 48 hours; have a current presence of vulvar, anal and or vaginal genital warts.
* Have had vaginal intercourse with a male partner within the last 48 hours.
* Current tobacco use.
* Are currently participating in another research study.

ELIGIBILITY:
Inclusion Criteria:

* Be of age 18 - 50 years-old, inclusive;
* Have a current BV infection (Nugent score 7 - 10) or intermediate vaginal flora (Nugent score 4 - 6), as diagnosed by Nugent score in the clinic (with later validation of the Nugent score by a blinded separate laboratory);63
* Regular menses with the last 2 menses 21-35 days apart;
* Willing and able to comply with study procedures, including the use of oral treatment for BV.

Exclusion Criteria:

* Contraindications to the use of oral metronidazole including:

  * Daily alcohol consumption and be unable or unwilling to abstain from alcohol while taking metronidazole tablets;
  * Known hypersensitivity to oral metronidazole;
* Chronic immune suppression (including, but not limited to chronic steroid use, chronic anti-fungal use, Diabetes Mellitus, organ transplant);
* An abnormal Pap smear documented in the past 12 months defined as:

  * ASC-US without a normal repeat Pap smear at least 6 months later;
  * ASC-US with positive reflex high-risk HPV testing (ASC-US/HPV+), low grade squamous epithelial lesion or high grade squamous intraepithelial lesion, ASC-H, atypical glandular cells, or malignant cells;
* It has been less than 3 months since the patient's last Depo medroxyprogesterone acetate (DMPA) injection and she has not had 2 normal, spontaneous menses since last using DMPA;
* Use of any other hormonal contraceptive method within past 2 months (oral, transdermal, transvaginal, implant, or hormonal intrauterine device);
* Use of oral or vaginal antibiotics or anti-fungals in the last 14 days;
* Surgery or biopsy of the vulva, vagina, or cervix within the past 30 days;
* History of hysterectomy;
* Pregnancy within the past 3 months;
* Current breastfeeding;
* HIV-1 sero-positivity in the participant (by history or buccal HIV-1 swab) or her current sexual partner(s);
* Current use of anti-viral suppression medications for Herpes Simplex Virus (HSV) (a history of HSV without active lesions is permitted);
* Current active sexually transmitted infection (STI);
* Presence of vaginal semen in the last 48 hours, per patient's report or as detected by prostate specific antigen (PSA) test;
* Use of douches, vaginal products or anything in the vagina in the past 48 hours;
* Current presence of vulvar, anal and or vaginal genital warts;
* Current tobacco use (any amount)
* Other conditions that, in the opinion of the investigator, would constitute contraindications to participation in the study or would compromise ability to comply with the study protocol, such as any major chronic illness including cancer, serious autoimmune disease or a major psychiatric disorder not under good control; and
* Current participation in any other drug or device study, or any study which, in the opinion of the investigator, would jeopardize interpretation of results of this study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea R Thurman, MD, Principal Investigator — CONRAD Eastern Virginia Medical School
Locations (1):
- Eastern Virginia Medical School CONRAD Clinical Research Center, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Cohort data will be published but not IPD

REFERENCES:
- [Derived] Gustin AT, Thurman AR, Chandra N, Schifanella L, Alcaide M, Fichorova R, Doncel GF, Gale M Jr, Klatt NR. Recurrent bacterial vaginosis following metronidazole treatment is associated with microbiota richness at diagnosis. Am J Obstet Gynecol. 2022 Feb;226(2):225.e1-225.e15. doi: 10.1016/j.ajog.2021.09.018. Epub 2021 Sep 22. PMID 34560047
- See also: CONRAD Reproductive Health — http://conrad.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for 6 months
Groups:
- Metronidazole: Open Label Study
Period: Overall Study
Arm/Group | Metronidazole
Started | 35
Completed | 33
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Metronidazole
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: p24 Antigen Production in Tissue
Description: The study will evaluate HIV infection and safety of cervico-vaginal tissue in women at 3 different time periods:
  1. During a BV infection
  2. Approximately 1 week after completing a 7-day course of metronidazole therapy
  3. Approximately 1 month after completing the 7-day course of metronidazole therapy
  Each of the 33 participants were sampled at baseline (during BV infection), approximately 1 week after treatment and approximately 1 month after treatment. p 24 antigen data was not evaluable in this study due to the fact that the samples were frozen prior to laboratory analyses, which damaged the samples. No data were collected.
Time Frame: 6 weeks
Arm/Group | Metronidazole
Number analyzed (Participants) | 0

2. Primary Outcome: p24 Antigen Production at Baseline Versus After Treatment With Metronidazole
Description: p 24 antigen data was not evaluable in this study due to the fact that the samples were frozen prior to laboratory analyses.
Time Frame: 30 days
Arm/Group | Metronidazole
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Metronidazole
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 2/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metronidazole (N=35)
Nausea (Gastrointestinal disorders) | 2 (2) — Nausea is commonly associated with metronidazole treatment

LIMITATIONS AND CAVEATS:
There were no serious adverse events related to product or procedures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No